CLINICAL TRIAL: NCT01238601
Title: Breast Implant Shell Geometry and Edge Scalloping: A Study Using the Upright MRI Machine
Brief Title: Upright Magnetic Resonance Imaging (MRI) Study - Breast Implant Shell Geometry and Edge Scalloping
Status: Completed | Type: Observational
Sponsor: Ideal Implant Incorporated (Industry)
Responsible Party: Robert S Hamas, MD, President, Ideal Implant Incorporated
Other Study IDs: Imaging Study of Implants
Record Dates: First submitted 2010-11-09; First posted 2010-11-10 (Estimated); Last update posted 2010-11-11 (Estimated); Status verified 2010-11

CONDITIONS: Breast Augmentation
Keywords: Breast augmentation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

SUMMARY:
The purpose of this study is to determine how different types of breast implants contour to the chest wall.

ELIGIBILITY:
Inclusion Criteria:

* had previous primary breast augmentation
* had previous replacement of breast implants
* has Baker Class I breast implant capsule

Exclusion Criteria:

* has scar capsule contracture around the breast implants of Baker Class II-IV
* is pregnant or may be pregnant
* has possibility or previous history of metallic foreign body

Ages: 20 Years to 50 Years | Sex: Female
Age Groups: Adult
Study Population: Women 20-50 who previously had primary breast augmentation or replacement of existing breast implants.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2007-07; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)